CLINICAL TRIAL: NCT04893096
Title: Rescue Therapy with the Human Anti-CD38 Antibody MOR202 (felzartamab) in Patients with Membranous Nephropathy Who Failed Anti-CD20 Target Therapy
Brief Title: MOR202 for Refractory MN
Acronym: MONET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: MorphoSys AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MONET; 2021-000835-30 (EudraCT Number)
Record Dates: First submitted 2021-05-11; First posted 2021-05-19 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Membranous Nephropathy
Keywords: membranous nephropathy; Anti-CD38; MOR 202
MeSH Terms: conditions — Glomerulonephritis, Membranous | interventions — felzartamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MOR202 (felzartamab) infusion (Experimental): Participants will receive active treatment for a total of nine doses during 24 weeks.
  Interventions: Drug: MOR202

INTERVENTIONS:
Drug: MOR202 — Each patient will be treated for 24 weeks and received a total of 9 doses. During the first treatment cycle, MOR202 will be administered weekly. For the following 5 months, patients will receive one dose every 4 weeks.
  Other Names: FELZARTAMAB

SUMMARY:
Membranous nephropathy (MN) - the leading cause of nephrotic syndrome (NS) in adults - is an immune-mediated disease that results from the deposition of immunoglobulins and complement components onto the sub-epithelial layer of the glomerular capillary wall. The availability for clinical use of rituximab, a monoclonal antibody against the B-cell surface antigen CD20, offered the opportunity to test the effects of specific CD20-targeted intervention aimed to prevent B-cell dependent mechanisms resulting in the production of nephritogenic autoantibodies. Rituximab-induced B-cell depletion reduced proteinuria in eight patients with MN while avoiding the adverse effects of steroids and other immunosuppressants. Subsequent studies confirmed that rituximab is remarkably safer than non-specific immunosuppressive agents, including cyclosporine, and achieves remission in approximately two-thirds of patients with MN-associated nephrotic syndrome. After rituximab-induced remission, however, NS may relapse in approximately one third of patients. Thus, novel therapeutic options are needed for a substantial proportion of patients with MN who may fail rituximab therapy. Conceivably, in patients with MN refractory to CD20-targeted therapy, the production of nephritogenic autoantibodies is sustained by mechanisms that do not depend on autoreactive CD20+ B cells.

Recently, it was shown that CD19-negative bone marrow plasma cells, which express CD38, are enriched in chronically inflamed tissue and secrete autoantibodies. Treatment of patients with MN with CD38-targeting antibodies may represent a new therapeutic approach.

MOR202 is a fully human recombinant monoclonal antibody against CD38 that has demonstrated in-vitro and in-vivo efficacy in experimental models of multiple myeloma. Antibody-dependent cellular cytotoxicity and antibody-dependent cellular phagocytosis are the principal mechanisms of action for MOR202-induced lysis of myeloma cells.

The working hypothesis is that CD38-targeted therapy with MOR202 may abrogate autoantibody-dependent mechanisms in patients with plasma-cell mediated forms of MN who failed previous treatment with rituximab and second-generation anti-CD20 monoclonal antibodies such as ofatumumab. With this background, MOR202 therapy may have an indication for patients with MN and NS resistant to CD20 targeted therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Biopsy-proven membranous nephropathy with or without detectable circulating anti-PLA2R or anti-THSD7A antibodies.
* Background treatment with RAS blocking agents (ACE inhibitor and/or ARBs), at maximum tolerated doses and adequately controlled blood pressure (BP <140/90 mmHg in at least three consecutive readings at screening).
* One condition between:
* Anti-CD20 Resistance: residual proteinuria ≥3.5 g/day (mean of three consecutive 24-hour urine collections), with less than 50% reduction compared to pre-treatment values at least 12 months after anti-CD20 antibody therapy.
* Anti-CD20 Dependence: frequently relapsing NS (nephrotic-range proteinuria for >50% of time in the last five years or since disease onset, whichever is shorter) despite repeated treatments with anti-CD20 antibodies.
* Estimated GFR >30 ml/min/1.73m2 (CKD-EPI equation) and less than 50% of sclerotic glomeruli in patients receiving renal biopsy.
* A minimum 12-month wash-out from last anti-CD20 therapy with rituximab and/or other monoclonal antibodies.
* No significant (i.e. more than 2 weeks) immunosuppressive therapy over the last 6 months.
* Written informed consent.

Exclusion Criteria:

* Clinically relevant neutropenia (neutrophils < 1.5 x 109/L), anemia (Hb levels <9.0 g/dL), thrombocytopenia (platelet count < 150.000/mm3), increased liver transaminase or bilirubin levels (total bilirubin, aspartate aminotransferase or alanine aminotransferase >1.5 x ULN, alkaline phosphatase >3.0 x ULN).
* Significant uncontrolled cardiovascular disease (including arterial or venous thrombotic or embolic events over the last three months) or cardiac insufficiency (New York Heart Association [NYHA] class IV) as judged by the investigator.
* Clinically relevant findings on a 12-lead electrocardiogram (ECG) as determined by the investigator at screening.
* History of significant cerebrovascular disease (stroke or transitory ischemic attack over the last three months) or sensory or motor neuropathy of toxicity ≥ grade 3.
* Any clinical condition that in the investigator judgment could affect the possibility to complete the study or could have a major confounding effect on study findings and data interpretation.
* Known intolerance to the study drug or its excipients
* Any viral, bacterial or fungal infection without complete symptoms resolution from at least two weeks.
* Serologic or virologic markers positive for HIV, hepatitis C (patients with positive antihepatitis C virus [anti-HCV] antibody but negative HCV RNA polymerase chain reaction [PCR] can enroll) or active or latent hepatitis B (patients with positive hepatitis B surface antigen [HBsAg] are excluded). Patients with isolated positive hepatitis B core antibody [anti-HBc], hepatitis B virus (HBV) DNA test by PCR must be non-detectable to enroll.
* History of malignancy within the prior 5 years.
* Participation in other clinical trials within 4 weeks of signing the consent form.
* Expected need of anti SARS Cov 2 vaccination during the study period
* Pregnancy or breast-feeding.
* Childbearing potential in males and females non using an highly effective method of contraception according to 2020 CTFG Recommendations related to contraception and pregnancy testing in clinical trials (https://www.hma.eu/fileadmin/dateien/Human_Medicines/01-About_HMA/Working_Groups/CTFG/2020_09_HMA_CTFG_Contraception_guidance_Version_1.1_updated.pdf).
* Legal incapacity or limited legal capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2025-02-21 (Actual); Study Completion 2025-02-21 (Actual)

PRIMARY OUTCOMES:
Change in 24-hour urinary protein excretion | Changes from screening and baseline, 1, 5,6,9,12,18 and 24 months after the first MOR202 administration.
Complete remission or partial remission of nephrotic syndrome. | Changes from screening and baseline, 1, 5,6,9,12,18 and 24 months after the first MOR202 administration.
  Complete remission is intended as : 24-hour urinary protein excretion <0.3 g or urinary protein to creatinine ratio < 300 mg/g, with serum albumin > 3.5 g/dL.
  Partial remission is intended as: 24-hour urinary protein excretion <3.5 g or urinary protein to creatinine ratio < 3500 mg/g, with at least 50% reduction compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Remuzzi, MD, Study Director — Istituto Di Ricerche Farmacologiche Mario Negri
Locations (2):
- Italy (2):
  - ASST HPG23 - Unità di Nefrologia, Bergamo, BG
  - Centro di Ricerche Cliniche per le Malattie Rare "Aldo e Cele Daccò", Ranica, BG